CLINICAL TRIAL: NCT06966154
Title: A Phase Ib/II Clinical Study Evaluating the Safety and Efficacy of Tislelizumab in Combination With Golidocitinib and Selinexor for the Treatment of Relapsed/Refractory Natural Killer/T-Cell Lymphoma (NKTCL)
Brief Title: A Phase Ib/II Clinical Study Evaluating the Safety and Efficacy of Tislelizumab in Combination With Golidocitinib and Selinexor for the Treatment of R/R NKTCL
Status: Recruiting | Phase: Phase 1 / Phase 2 | Type: Interventional
Sponsor: Fudan University (Other)
Responsible Party: Principal Investigator, Rong Tao, Professor & Chief, Fudan University
Allocation: Randomized | Model: Sequential | Masking: None | Purpose: Treatment
Other Study IDs: SHCA-NKT-202501
Record Dates: First submitted 2025-05-02; First posted 2025-05-11 (Actual); Last update posted 2025-05-30 (Actual); Status verified 2025-05

CONDITIONS: Natural Killer/T-cell Lymphoma; Relapsed or Refractory Lymphoma Including ENKL
Keywords: natural killer/T-cell lymphoma; Immune checkpointor inhibitor; tislelizumab; golidocitinib; selinexor
MeSH Terms: conditions — Recurrence | interventions — selinexor

STUDY DESIGN:
Intervention Model Description: Phase Ib (Safety Run-In Section) Guided by the Bayesian Optimal Interval (BOIN) design, the study explores the combined dosing of golidocitinib, selinexor, and tislelizumab across 2 dose levels and 4 dosing cohorts . Patients are sequentially enrolled in chronological order and assigned to one of the following combination regimens: Golidocitinib: 2 dose groups. Selinexor: 2 dose groups.Randomization is implemented within each dose level. The first treatment cycle (28-day cycle) is designated as the dose-limiting toxicity (DLT) observation period.
  Dose Escalation Rules:
  If both cohorts at Dose Level 1 (golidocitinib + selinexor combinations) demonstrate acceptable tolerability per the SRC, golidocitinib is escalated to the higher dose in Dose Level 2.
  If either cohort at Dose Level 1 is deemed intolerable by the SRC, de-escalation to Dose Level 0 (baseline dose) is mandated.
  Following completion of all 4 cohorts in Phase Ib, the recommended dose (RP2D) will be determined.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (1):
- tislezumab plus golidocitinib and selinexor (Experimental): Patients will receive Tislelizumab: Fixed intravenous dose of 200 mg every 3 weeks (Q3W).
  Golidocitinib: Dose-escalating oral regimens:
  Dose level A: 150 mg every other day (QOD). Dose level B: 150 mg once daily (QD).
  Selinexor: Dose-escalating oral regimens:
  Dose A: 40 mg once weekly (QW) . Dose B: 60 mg QW for 2 consecutive weeks, followed by 1 week off. Safety monitoring will be performed throughout each 3-week cycle, with dose escalation contingent on safety/tolerability assessments.
  Interventions: Drug: tislezumab; Drug: golidocitinib; Drug: Selinexor

INTERVENTIONS:
Drug: tislezumab — Tislelizumab will be administered intravenously at a fixed dose of 200 mg every 3 weeks (Q3W).
Drug: golidocitinib — Golidocitinib: Dose-escalating oral regimens:
  Dose level A: 150 mg every other day (QOD). Dose level B: 150 mg once daily (QD).
Drug: Selinexor — Selinexor: Dose-escalating oral regimens: Dose A: 40 mg once weekly (QW) . Dose B: 60 mg QW for 2 consecutive weeks, followed by 1 week off.

SUMMARY:
This open-label, multicenter Ib/II phase clinical trial investigates the safety, tolerability, and preliminary efficacy of tislezumab (anti-PD-1 monoclonal antibody), golidocitinib (JAK1/STAT3 signaling pathway inhibitor), and selinexor (selective inhibitor of nuclear export, XPO1 antagonist) in patients with relapsed/refractory extranodal natural killer/T-cell lymphoma (R/R ENKTL) progressing after ≥1 line of L-asparaginase-containing chemotherapy or chemoradiotherapy.

DETAILED DESCRIPTION:
This phase Ib/II open-label, multicenter clinical trial addresses the critical unmet need in relapsed/refractory extranodal natural killer/T-cell lymphoma (R/R ENKTL), an aggressive Epstein-Barr virus (EBV)-associated non-Hodgkin lymphoma subtype characterized by extranodal predominance, angiocentric growth patterns, and geographic prevalence in Asian and Latin American populations. Despite incorporation of L-asparaginase-based regimens into first-line therapy, approximately 30-40% of patients experience primary refractory disease or relapse, with median overall survival (OS) of <6 months in PD-1 inhibitor-resistant cohorts and limited sustained responses to salvage therapies, highlighting the imperative for novel mechanism-driven combinations. The investigational triplet regimen-comprising tislelizumab (anti-PD-1 monoclonal antibody), golidocitinib (JAK1/STAT3 inhibitor), and selinexor (XPO1 antagonist)-was rationally designed to exploit synergistic mechanisms targeting ENKTL pathogenesis: PD-1 blockade reverses T-cell exhaustion, JAK/STAT3 inhibition disrupts constitutive oncogenic signaling (e.g., STAT3 Y705 phosphorylation), and XPO1 antagonism promotes nuclear retention of tumor suppressors (p53, IkBα) while destabilizing EBV latency proteins. Part 1 (Phase Ib) employs dose escalation across combinatorial cohorts to establish the recommended Phase II dose (RP2D), prioritizing safety and tolerability through rigorous assessment of dose-limiting toxicities (DLTs), while Part 2 (Phase II) evaluates preliminary efficacy in a dedicated anti-PD-1-refractory population, focusing on objective response rate (ORR) by Lugano 2014 criteria as the primary endpoint. The trial specifically targets patients with histologically confirmed ENKTL per WHO classification and radiographically confirmed progression post-L-asparaginase-containing therapy and failed to prior anti-PD-1/PD-L1 therapy, excluding those with prior exposure to JAK or XPO1 inhibitors to isolate the novel therapeutic effect. By integrating PD-1 pathway modulation with simultaneous disruption of STAT3-driven survival signals and viral oncoprotein dependencies, this combination strategy aims to discover the potential therapeutic paradigms for R/R ENKTL, particularly in populations failing contemporary immunochemotherapy approaches.

ELIGIBILITY:
Inclusion Criteria:

* Voluntarily participate in the clinical study; fully understand and provide informed consent (via a signed Informed Consent Form, ICF); willing and able to comply with all trial procedures.
* Histopathologically confirmed diagnosis of extranodal NK/T-cell lymphoma, nasal type (NKTCL) by the participating study center.
* Relapsed or refractory NKTCL after failure of asparaginase-based chemotherapy ± radiotherapy:

  * Relapse: Disease recurrence >6 months after achieving complete response (CR) to prior therapy.
  * Refractory: Failure to achieve CR or disease progression after adequate systemic therapy (≥4 cycles of a combination regimen).
  * For Phase II: Patients must have received prior anti-PD-1 monoclonal antibody therapy and remain refractory.
* At least one measurable or evaluable lesion per Lugano 2014 criteria:

  * Measurable lesion: CT/MRI: Longest diameter ≥1.5 cm (lymph nodes) or ≥1.0 cm (extranodal lesions).Post-radiation lesions require radiological evidence of progression.
  * Evaluable lesion: FDG-PET: Lymph node/extranodal lesion with uptake > liver and imaging consistent with lymphoma.
* Age ≥18 years at the time of ICF signing.
* Life expectancy >12 weeks.
* ECOG performance status 0-2.
* Adequate organ and bone marrow function:

  * Hematology (no transfusion/G-CSF support within 14 days): ANC ≥1.5×10⁹/L (≥0.5×10⁹/L if bone marrow involvement)；Platelets ≥100×10⁹/L (≥50×10⁹/L if bone marrow involvement)；Hemoglobin ≥8.0 g/dL.
  * Liver function: Total bilirubin ≤1.5×ULN (≤3.0×ULN for Gilbert's syndrome or liver involvement).

ALT/AST ≤2.5×ULN (≤5.0×ULN with liver involvement).

* Renal function: Serum creatinine ≤1.5×ULN OR creatinine clearance (Cockcroft-Gault) ≥50 mL/min.
* Coagulation: INR ≤1.5×ULN; PT/APTT ≤1.5×ULN (unless on anticoagulants within therapeutic range).
* Cardiac function: LVEF ≥50% by echocardiography (ECHO).

  * Recovery from prior anticancer therapy toxicities to CTCAE v5.0 Grade ≤1 or baseline. Exceptions: Irreversible Grade 2 toxicities unlikely to worsen during the study (e.g., neuropathy, alopecia) per investigator's assessment.
  * For women of childbearing potential (WOCBP): Negative serum pregnancy test within 7 days before enrollment. WOCBP and male participants with WOCBP partners must agree to use effective contraception from ICF signing until ≥6 months after the last study dose.

Exclusion Criteria:

* History of malignancy within the past 5 years, with the exception of: Locally curable malignancies treated with curative intent (e.g., basal or squamous cell skin cancer, thyroid carcinoma, superficial bladder cancer, or in situ carcinoma of the prostate, cervix, or breast).
* Any of the following prior treatments:

  * History of allogeneic hematopoietic stem cell transplantation (allo-HSCT) within 5 years prior to the first dose (patients with allo-HSCT >5 years before the first dose and no active graft-versus-host disease may enroll).
  * Autologous hematopoietic stem cell transplantation (auto-HSCT) within 3 months prior to the first dose.
  * Prior use of JAK inhibitors, STAT3 inhibitors, or XPO1 inhibitors.
  * Current use of vitamin K antagonists, antiplatelet agents, or anticoagulants (or inability to discontinue within 1 week before the first dose).
  * Systemic glucocorticoids or immunosuppressants within 14 days prior to enrollment (allowed: topical, ocular, intra-articular, intranasal, or inhaled glucocorticoids; short-term [≤7 days] prophylactic use for non-autoimmune conditions).
  * Cytotoxic chemotherapy within 14 days prior to enrollment.
  * Systemic anticancer therapy (including monoclonal antibodies or immunotherapy) within 4 weeks prior to the first dose.
  * Major organ surgery within 6 weeks or radiotherapy within 90 days prior to enrollment.
  * Radioimmunoconjugate therapy within 10 weeks prior to enrollment.
  * Use of other investigational drugs requiring investigator's risk-benefit assessment.
  * Participation in other clinical trials with investigational drugs within 30 days prior to enrollment.
  * Vaccines (except influenza vaccines) within 28 days prior to enrollment.
* Active infections, including:

  * Active or latent tuberculosis (positive tuberculin skin test [PPD] with induration ≥10 mm or radiologically confirmed active lesions).
  * Known HIV infection or AIDS.
  * Chronic active hepatitis B or C:

HBV: Exclude if HBV DNA detectable (↑center-specific ULN). HCV: Exclude if HCV RNA detectable (↑center-specific ULN).

* Other active viral infections (e.g., herpes zoster, CMV) requiring treatment. Infections requiring intravenous antimicrobial therapy.

  * Uncontrolled cardiac conditions, including:
* NYHA Class >II heart failure.
* Unstable angina.
* Myocardial infarction within 1 year.
* Clinically significant arrhythmias requiring intervention.

  * Persistent drug-related toxicities >CTCAE Grade 1 (excluding alopecia) at baseline.
  * Uncontrolled nausea/vomiting, chronic gastrointestinal diseases, dysphagia, or prior bowel resection affecting drug absorption.
  * Pregnancy, lactation, or refusal to use contraception by participants of reproductive potential.
  * Psychiatric disorders or inability to provide informed consent.
  * Other conditions deemed unsuitable for study participation by the investigator.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 68 (Estimated)
Dates: Start 2025-05-26 (Actual); Primary Completion 2027-05-30 (Estimated); Study Completion 2028-05-30 (Estimated)

PRIMARY OUTCOMES:
RP2D of golidocitinib in combination with selinexor | 4 weeks after the initiation of combination treatment
  Recommended Phase II Dose of golidocitinib in combination with selinexor
Satety profile | 6 months after the last lose of combination treatment
  Safety profile, including: Incidence, severity, and drug-relatedness of adverse events (AEs) and serious adverse events (SAEs) per NCI CTCAE ver 5.0
Overall response rate | 12-weeks after the initiation of combination treatment
  Phase II (Dose-Expansion Phase) part 12-week objective response rate (ORR) assessed per Lugano 2014 criteria for lymphoma response evaluation.

SECONDARY OUTCOMES:
Complete Response Rate | 12-weeks after the initiation of combination treatment
  Phase II (Dose-Expansion Phase) part 12-week complete response rate (CRR) assessed per Lugano 2014 criteria for lymphoma response evaluation.
Duration of Response | 12 months after the last patient enrolled
  Duration of Response (DoR) per Lugano 2014 response criteria
Progression-Free Survival (PFS) | 12 months after the last patient enrolled
  The length of time from the start of treatment until disease progression or death from any cause, whichever occurs first.
Overall survival(OS) | 12 months after the last patient enrolled
  The length of time from the start of treatment until death from any cause.
Treatment-Emergent Adverse Events（TEAE） | 6 months after the last patient quit the trial treatment
  The incidence of TEAEs (Treatment-Emergent Adverse Events), AEs/SAEs/immune-related adverse events (irAEs), their association with the investigational drug, and their severity as assessed according to CTCAE v5.0.

OTHER OUTCOMES:
Biomarkers | 6 months after the last patient enrolled
  Predictive Biomarkers of Treatment Efficacy and safety

CONTACTS AND LOCATIONS:
Locations (1):
- Dept of lymphoma and medical oncology, Shanghai Cancer Center, Shanghai, Shangai, China

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Background] Kwong YL, Chan TSY, Tan D, Kim SJ, Poon LM, Mow B, Khong PL, Loong F, Au-Yeung R, Iqbal J, Phipps C, Tse E. PD1 blockade with pembrolizumab is highly effective in relapsed or refractory NK/T-cell lymphoma failing l-asparaginase. Blood. 2017 Apr 27;129(17):2437-2442. doi: 10.1182/blood-2016-12-756841. Epub 2017 Feb 10. PMID 28188133
- [Background] Tao R, Liu C, Zhang W, Zhu Y, Ma Y, Hao S. Selinexor With Anti-PD-1 Antibody as a Potentially Effective Regimen for Patients With Natural Killer/T-Cell Lymphoma Failing Prior L-Asparaginase and PD-1 Blockade. Oncologist. 2024 Jan 5;29(1):e90-e96. doi: 10.1093/oncolo/oyad241. PMID 37616529
- [Background] Mathew D, Marmarelis ME, Foley C, Bauml JM, Ye D, Ghinnagow R, Ngiow SF, Klapholz M, Jun S, Zhang Z, Zorc R, Davis CW, Diehn M, Giles JR, Huang AC, Hwang WT, Zhang NR, Schoenfeld AJ, Carpenter EL, Langer CJ, Wherry EJ, Minn AJ. Combined JAK inhibition and PD-1 immunotherapy for non-small cell lung cancer patients. Science. 2024 Jun 21;384(6702):eadf1329. doi: 10.1126/science.adf1329. Epub 2024 Jun 21. PMID 38900877
- [Background] Song Y, Malpica L, Cai Q, Zhao W, Zhou K, Wu J, Zhang H, Mehta-Shah N, Ding K, Liu Y, Li Z, Zhang L, Zheng M, Jin J, Yang H, Shuang Y, Yoon DH, Gao S, Li W, Zhai Z, Zou L, Xi Y, Koh Y, Li F, Prince M, Zhou H, Lin L, Liu H, Allen P, Roncolato F, Yang Z, Kim WS, Zhu J. Golidocitinib, a selective JAK1 tyrosine-kinase inhibitor, in patients with refractory or relapsed peripheral T-cell lymphoma (JACKPOT8 Part B): a single-arm, multinational, phase 2 study. Lancet Oncol. 2024 Jan;25(1):117-125. doi: 10.1016/S1470-2045(23)00589-2. Epub 2023 Dec 9. PMID 38092009
- [Background] Tao R, Fan L, Song Y, Hu Y, Zhang W, Wang Y, Xu W, Li J. Sintilimab for relapsed/refractory extranodal NK/T cell lymphoma: a multicenter, single-arm, phase 2 trial (ORIENT-4). Signal Transduct Target Ther. 2021 Oct 27;6(1):365. doi: 10.1038/s41392-021-00768-0. PMID 34702811